CLINICAL TRIAL: NCT03806088
Title: Prevalence of Electrolyte Imbalance in Chronic Kidney Disease: A Study at Tertiary Care Hospitals in South Punjab, Pakistan
Brief Title: Prevalence of Electrolyte Imbalance in Chronic Kidney Disease:A Study at Tertiary Care Hospital in South Punjab,Pakistan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Hafiz Muhammad Attaullah, HAFIZ MUHAMMAD ATTAULLAH student of pharm-D, Islamia University of Bahawalpur
Other Study IDs: IslamiaUS
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Chronic Kidney Diseases
Keywords: CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients of chronic kidney disease: no interventions

SUMMARY:
an observational cross-sectional study is done to calculate the electrolyte imbalance at different stages of chronic kidney disease at tertiary care hospital.

DETAILED DESCRIPTION:
an observational cross-sectional study is done to calculate the electrolyte imbalance at different stages of chronic kidney disease at tertiary care hospitals of south Punjab, Pakistan .The outcomes of chronic kidney disease and end stage of renal failure will be calculated according to standard protocol. Under the supervision of pathologists, pharmacologists, pharmacists, nephrologists, urologists and biostatistician. The standard protocol was authorized by ethical committee of each center. patient consent form was

ELIGIBILITY:
Inclusion Criteria:

* CKD patients ranging
* age from 20-80
* dialysis and pre-dialysis patients
* who provide written consent form

Exclusion Criteria:

* congenital one kidney patients
* organ or kidney donors and transplantation
* pregnant women
* renal injury during trauma

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An observational cross sectional study is done on pakistani population while working in different tertiary care hospitals of south Punjab including Bahawal Victoria hospital Bahawalpur, kidney center Multan and many registered clinics, under the supervision of pathologists, pharmacologists,pharmacists,nephrologists,urologists and biostatistician.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Estimated)

PRIMARY OUTCOMES:
Serum potassium in mEq/L | 2days
  Serum potassium in mEq/L by taking blood sample under standard condition
serum urea in mg/dl | 2days
  serum urea in mg/dl by taking blood sample under standard condition
Serum creatinine in mg/dl | 2days
  Serum creatinine in mg/dl by taking blood sample under standard condition
Serum calcium in mg/dl | 2days
  Serum calcium in mg/dl by taking blood sample under standard condition
Serum sodium in mEq/L | 2days
  Serum sodium in mEq/L by taking blood sample under standard condition

SECONDARY OUTCOMES:
Blood pressure in mm of Hg | 2days
  Blood pressure in mm of Hg
Blood glucose concentration in mg/dl | 2days
  Blood glucose concentration in mg/dl random

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy and Alternative Medicine Khawaja Freed Campus, Chak Four Hundred Fifty-four, Punjab Province, Pakistan